CLINICAL TRIAL: NCT03782662
Title: An Adaptive, Part Open-label, Part Randomised Phase 1 Clinical Trial in Healthy Volunteers to Study Drug Interactions With RV521 Including Those Mediated by CYP3A4 and P-glycoprotein
Brief Title: A Study to Learn About the Drug-drug Interactions of Sisunatovir in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: REVC004; C5241004 (Other: Alias Study Number); 2018-003256-21 (EudraCT Number)
Record Dates: First submitted 2018-12-05; First posted 2018-12-20 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Itraconazole; Verapamil; Rifampin; Midazolam; sisunatovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- RV521 plus Itraconazole (Experimental): RV521 drug substance in capsule for oral administration, a single 200 mg dose administered on D1 and a single 200 mg dose administered on D7 plus Itraconazole 100 mg capsules for oral administration, a 200 mg dose administered once daily on D4 - D10, inclusive
  Interventions: Drug: Itraconazole; Drug: RV521
- RV521 plus Verapamil (Experimental): RV521 drug substance in capsule for oral administration, a single 200 mg dose administered on D1 and a single 200 mg dose administered on D11 plus Verapamil, 80 mg tablets for oral administration, an 80 mg dose administered TDS daily on D4 - D14, inclusive
  Interventions: Drug: Verapamil; Drug: RV521
- RV521 plus Rifampicin (Experimental): RV521 drug substance in capsule for oral administration, a single 200 mg dose administered on D1 and a single 200 mg dose administered on D10 plus Rifadin, Rifampicin, 300 mg capsules for oral administration, a 600 mg dose administered once daily on D4 - D10, inclusive
  Interventions: Drug: Rifampicin; Drug: RV521
- RV521 plus Midazolam (Experimental): RV521 drug substance in capsule for oral administration, 200 mg dose administered BID on D2 - D15, inclusive plus Buccolam 10 mg oromucosal solution of midazolam, oral syringes, a single 10 mg dose administered on D1 and a single 200 mg dose administered on D15
  Interventions: Drug: Midazolam; Drug: RV521
- Placebo plus Midazolam (Placebo Comparator): Placebo for RV521 in capsule for oral administration, 200 mg dose administered BID on D2 - D15, inclusive plus Buccolam 10 mg oromucosal solution of midazolam, oral syringes, a single 10 mg dose administered on D1 and a single 200 mg dose administered on D15
  Interventions: Drug: Midazolam; Drug: Placebo for RV521

INTERVENTIONS:
Drug: Itraconazole — Itraconazole capsules
  Arms: RV521 plus Itraconazole
Drug: Verapamil — Verapamil tablets
  Arms: RV521 plus Verapamil
Drug: Rifampicin — Rifampicin capsules
  Other Names: Rifadin
  Arms: RV521 plus Rifampicin
Drug: Midazolam — Midazolam oromucosal solution
  Other Names: Midazolam Prefilled Syringe; Buccolam
  Arms: Placebo plus Midazolam; RV521 plus Midazolam
Drug: Placebo for RV521 — Placebo for RV521 capsules
  Arms: Placebo plus Midazolam
Drug: RV521 — RV521 capsules
  Arms: RV521 plus Itraconazole; RV521 plus Midazolam; RV521 plus Rifampicin; RV521 plus Verapamil

SUMMARY:
The purpose of this clinical trial is to learn about the interaction of sisunatovir with four medications (midazolam, itraconazole, rifampicin, and verapamil). These medications are known to have specific effects on enzymes and proteins that could influence drug absorption.

This study will be conducted in 4 Cohorts:

* Cohort 1 will receive midazolam and sisunatovir or placebo,
* Cohort 2 will receive Itraconazole and sisunatovir,
* Cohort 3 will receive verapamil and sisunatovir,
* Cohort 4 will receive rifampicin and sisunatovir. A placebo looks like sisunatovir but does not contain any active medicine in it.

This study is looking for health adult participants that meet the following criteria:

1. Caucasians age 18 to 45 years
2. All fertile participants must agree to the use of highly effective contraception
3. Body mass index (BMI) of 18-25.0 kg/m2
4. Male and female participants who are overtly healthy as determined by medical evaluation. This includes medical history, physical examination, blood pressure, pulse rate, standard 12-lead ECG (electrocardiogram), and laboratory tests.

This study consists of 2 parts, Part A and Part B. Part A will enroll up to 104 participants. The design of Part B will be determined after the completion of Part A.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years, inclusive
* Willing to comply with protocol defined contraception requirements
* In good health with no history of major medical conditions
* A body mass index (BMI) of 18 - 25 kg/m2

Exclusion Criteria:

* Evidence of any clinically significant or currently active major medical condition
* Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab)
* Not willing to comply with protocol defined restrictions for intake of drugs of abuse, alcohol, nicotine-containing products, medication (prescription, OTC, herbal, vitamins/minerals etc) and specified food and drink products

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-03-17 (Actual)

PRIMARY OUTCOMES:
Effect of RV521 on Cmax of Midazolam | Baseline to study day 17
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of RV521 on tmax of Midazolam | Baseline to study day 17
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of RV521 on t1/2 of Midazolam | Baseline to study day 17
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of RV521 on AUC of Midazolam | Baseline to study day 17
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of RV521 on CL/F of Midazolam | Baseline to study day 17
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of itraconazole on Cmax of RV521 | Baseline to study day 12
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of itraconazole on tmax of RV521 | Baseline to study day 12
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of itraconazole on t1/2 of RV521 | Baseline to study day 12
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of itraconazole on AUC of RV521 | Baseline to study day 12
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of itraconazole on CL/F of RV521 | Baseline to study day 12
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of verapamil on Cmax of RV521 | Baseline to study day 16
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of verapamil on tmax of RV521 | Baseline to study day 16
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of verapamil on t1/2 of RV521 | Baseline to study day 16
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of verapamil on AUC of RV521 | Baseline to study day 16
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of verapamil on CL/F of RV521 | Baseline to study day 16
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of rifampicin on Cmax of RV521 | Baseline to study day 15
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of rifampicin on tmax of RV521 | Baseline to study day 15
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of rifampicin on t1/2 of RV521 | Baseline to study day 15
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of rifampicin on AUC of RV521 | Baseline to study day 15
  The specified pharmacokinetic parameter will be summarised using descriptive statistics
Effect of rifampicin on CL/F of RV521 | Baseline to study day 15
  The specified pharmacokinetic parameter will be summarised using descriptive statistics

SECONDARY OUTCOMES:
Number of subjects with treatment-related adverse events as assessed by NCI CTCAE V5.0 | Screening to final study visit (performed at 7 days following the last dose of any intervention)
  The number of subjects with treatment-related adverse events will be summarised by treatment group using descriptive statistics
Number of subjects with QT/QTc interval changes relative to baseline who received RV521 (monotherapy), Midazolam (monotherapy) or RV521 and Midazolam (combination therapy) | Baseline to to final study visit (performed at 7 days following the last dose of any intervention)
  Descriptive statistics will be given by time point and dose-group for absolute values and change from baseline. Results will be tabulated and for QTc, the difference to time matched placebo will also be displayed

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Richmond Pharmacology Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=REVC004